CLINICAL TRIAL: NCT05217680
Title: Phase III Non-inferiority Clinical Study to Evaluate the Efficacy and Safety of Intravitreous PRO-169 Compared to Ranibizumab for Diabetic Macular Edema
Brief Title: Clinical Study to Evaluate PRO-169 for Diabetic Macular Edema
Acronym: PRO-169
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH169-0718/III
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Intervention Model Description: Clinical study, phase III, multi-centric, randomized, double-blind, with active parallel control to show non-inferiority.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-169 (Experimental): Bevacizumab 1.25 mg / 0.05mL for intravitreal injection. All patients in this arm will be exposed to one monthly injection for the first four months. During the rest of the study, during the monthly visits, it will be decided if injections are to be continued or postponed. The maximum amount of intravitreal injections to be administered are 12.
  Interventions: Biological: Bevacizumab
- Lucentis ® (Active Comparator): Ranibizumab 0.5 mg / 0.05mL for intravitreal injection. All patients in this arm will be exposed to one monthly injection for the first four months. During the rest of the study, during the monthly visits, it will be decided if injections are to be continued or postponed. The maximum amount of intravitreal injections to be administered are 12.
  Interventions: Biological: Lucentis®

INTERVENTIONS:
Biological: Bevacizumab — Administration of monthly intravitreal bevacizumab (4-12 injections)
  Arms: PRO-169
Biological: Lucentis® — Administration of monthly intravitreal ranibizumab (4-12 injections)
  Arms: Lucentis ®

SUMMARY:
Phase III clinical study to evaluate the efficacy, expressed as improvement in visual acuity in patients suffering diabetic macular edema after one year of treatment with PRO-169, compared to treatment with Lucentis® (ranibizumab).

DETAILED DESCRIPTION:
A total of 442 patients with diabetic macular edema will be randomized 1:1 to be treated with either PRO-169 (bevacizumab) or Lucentis® (ranibizumab). There will be a total of 14 visits, including selection and final visits. Monthly evaluations will include ophthalmologic evaluations of anterior and posterior segments, as well as OCT (optic coherence tomography) to obtain central macular width and retinal volume. Fluorescein angiography will be performed on selection visit as well as 6 and 12 months into the study (visits 7 and 13). All patients will be exposed to intravitreal injection of either of the studied drugs monthly for the first 4 months. Starting on visit 5 patients will be injected depending on their response to treatment, calculated according predetermined algorithms including clinical and image variables. Starting on month 6, patients may be subjected to rescue therapy with photocoagulation if they comply with predetermined criteria for such measure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of Diabetes Mellitus (type 1 or 2) evidenced by: use of insulin or use of oral hypoglycemic medications or diagnosis for DM according to OMS or ADA criteria.
* Is capable of rendering informed consent.
* HbA1c <8.5% in selection visit.
* All men and women capable of reproduction may agree to use a barrier birth control method during the study and 3 months after the last intravitreal injection applied.
* Only one eye may be randomized per participating individual, in case both are eligible, the investigator may choose either eye according his/her criteria.
* BVCA according to ETDRS between <78 (20/32 or worse) and >24 (20/320 or better) within 8 days prior to the randomization.
* Clinically evident diabetic macular edema, with central macular thickening.
* Diabetic macular edema demonstrated in OCT scan (macular central thickness > 300 μm for men and > 290 μm for women) within 8 days prior to the randomization.
* Presenting characteristics that allow an adequate fundus examination (transparent means, adequate pupil dilation, etc).

Exclusion Criteria:

* Chronic renal disease with renal insufficiency that requires dialysis or transplant.
* Individuals with conditions that may compromise their participation during the span of the study (unstable concomitant diseases, possible change of residence, etc)
* Individuals with a poor glycemic control who have started insulin treatment within 4 months previous to the study.
* Participation in another clinical study (at least 90 days must have elapsed between the finalization of his/her participation in a previous essay and randomization in the present study).
* Known allergies to the treatment.
* Poorly controlled blood pressure (average of 3 readings while sitting with ≥160 mmHg systolic or ≥100 mmHg diastolic in the selection visit.
* Heart attack or other cardiovascular event (cerebral vascular disease, transitory ischemia, hospitalization for cardiac insufficiency) during the 4 months prior to the start of the study, or patients with active myocardial insufficiency.
* Previous systemic treatment with VEGF-related medications within 4 months prior to the start of the study.
* Women of child-bearing age who are pregnant, lactating of planning to get pregnant within the time span of the study.
* Known allergy to anesthetic medications used during the procedures, intravitreal injection and photocoagulation.
* Diagnosis of non-diabetic macular edema.
* Ophthalmic conditions that interfere with the evaluation of BCVA (for example: foveal atrophy, pigmentary abnormalities, dense foveal exudates, etc)
* Additional conditions to DM that may compromise the evaluation of the edema (for example: venous occlusions, uveitis or other inflammatory diseases, neovascular glaucoma, etc)
* Lens opacities that according to the LOCS III classification system exceed one or more of the following: > NO3C3, > C2, > P1.
* Previous history of anti-VEGF treatment for diabetic macular edema or any treatment for diabetic macular edema within 4 months prior to the start of the study (corticosteroids, photocoagulation, etc)
* Anticipation of the need of panphotocoagulation (for example: proliferative diabetic retinopathy or any other indication) during the period of the study or history of panphotocoagulation within the 4 months prior to the start of the study.
* History of ocular surgery (cataract extraction, any intraocular surgery, aphakia, etc) within 4 months prior to the start of the study, or planned to occur within the time span of the study.
* Intraocular pressure > 21 mmHg, measured through Goldmann tonometry during the selection visit.
* Presence of macular ischemia or important loss of perifoveal capilaries (avascular foveal zone greater than 350 μm) demonstrated through fluorescein angiography during the selection visit.
* Evidence of macular traction and hyaloid thickening in OCT scan.
* History of YAG capsulotomy within 2 months prior to the randomization.
* Evidence of external ocular infections or any important disease of the ocular surface.
* History of vitrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Best Corrected Visual Acuity will be evaluated according the standardized ETDRS. The mean change between two treatments will be used evaluated as difference between baseline and final (12 months) values.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity area under the curve | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Best Corrected Visual Acuity will be evaluated according the standardized ETDRS. The area under the curve of both treatments will be used evaluated as difference between baseline and final (12 months) values.
Best Corrected Visual Acuity (adjusted to baseline) | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5)
  Best Corrected Visual Acuity will be evaluated according the standardized ETDRS. The corrected BCVA (adjusted to baseline value) of both treatments will be used evaluated at 4 months.
Central Macular Thickness | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Central macular thickness will be evaluated through OCT scan. The mean change between two treatments will be used evaluated as difference between baseline and final (12 months) values.
Retinal Volume | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Retinal volume will be evaluated through OCT scan. The mean change between two treatments will be used evaluated as difference between baseline and final (12 months) values.
Percentage of patients with a positive response to treatment. | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Determining the percentage of patients with a positive response to treatment, considered as: absolute improvement (20/20 vision for two consecutive visits and central macular thickness < 300 μm in men and < 290 μm in women), improvement (one or more of the following: patient who gained 5 or more letters for BCVA, ≥ 10% decrease of macular central thickness value compared to last two visits) and stability (one or more of the following: patient with neither a gain of 5 or more letters for BCVA nor a ≥ 10% decrease of macular central thickness value compared to last two visits, patient without loss of 5 or more letters for BCVA or a ≥ 10% decrease of macular central thickness value compared to last visit).
Mean number of injections | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Determining the mean number of injections applied during study, comparing both arms.
Frequency of rescue therapy administration | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Determining the frequency of the need of photocoagulation as a rescue therapy, comparing in both arms.
Adverse Events | Days: 0 (selection), 1 (randomization), 30±3 (Visit 2), 60±3 (Visit 3), 90±3 (Visit 4), 120±3 (Visit 5), 150±3 (Visit 6), 180±3 (Visit 7), 210±3 (Visit 8), 240±3 (Visit 9), 270±3 (Visit 10), 300±3 (Visit 11), 330±3 (Visit 12), 360±3 (Final Visit)
  Determining the incidence and severity of adverse events presented during the study, comparing both arms in both systemic and ophthalmic adverse events (related to research products).

CONTACTS AND LOCATIONS:
Locations (2):
- Fundación Oftalmológica Nacional, Bogotá, Colombia
- SalaUno Salud, S.A.P.I. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salcedo-Villanueva G, Garcia-Sanchez G, Palacio-Pastrana C, Gascon-Guzman G, Moreno-Andrade A, Olvera-Montano O, Munoz-Villegas P. One-year results of visual response following intravitreal novel anti-VEGF injection for diabetic macular edema in a Latino population. Int J Retina Vitreous. 2025 Aug 1;11(1):89. doi: 10.1186/s40942-025-00719-9. PMID 40750915
- [Derived] Torres-Arellano JM, Tornero-Jimenez A, Sanchez-Rios A, Olvera-Montano O, Munoz-Villegas P. Evaluation of the Relationship Between Diabetic Macular Edema and Renal Function in a Latino Population. Ophthalmol Ther. 2023 Oct;12(5):2745-2755. doi: 10.1007/s40123-023-00787-w. Epub 2023 Aug 6. PMID 37543959